CLINICAL TRIAL: NCT03466021
Title: Effects of GLP-1 Receptor Agonist Treatment on Pulmonary Function and Quality of Life in Obese Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: Effects of Liraglutide in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Claus Bogh Juhl (Other)
Responsible Party: Sponsor-Investigator, Claus Bogh Juhl, MD. ph.d, Esbjerg Hospital - University Hospital of Southern Denmark
Organization: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1188-8695
Record Dates: First submitted 2018-03-02; First posted 2018-03-15 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GLP-1 receptor agonist; Chronic obstructive pulmonary disease; FDG/PET-CT; inflammation; weightloss; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation; Weight Loss | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, placebo-controlled, double-blinded, parallel group and two-center trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide (Active Comparator): Liraglutide injection 3.0 mg daily
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Placebo, matching injection pen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Initially 0.6 mg daily, increasing weekly with 0.6 mg, until 3.0 mg is reached.
  Other Names: Saxenda; NN2211
  Arms: Liraglutide
Drug: Placebo — Matching injection
  Arms: Placebo

SUMMARY:
The study is a 44 weeks, prospective, randomized, placebo-controlled, double-blinded, parallel group two-center trial. Forty patients are recruited among the outpatients of the chronic obstructive pulmonary disease (COPD) clinic, Hospital of South West Jutland and Lillebælt Hospital according to the inclusion and exclusion criteria. The patients are randomized to receive liraglutide 3 mg per day (initial dose 0.6 mg, increasing by 0.6 mg weekly until 3 mg is reached) or placebo. At baseline, after four weeks (assessment of the acute effect of liraglutide), 20 weeks, and 40 weeks (assessment of the combined effect of liraglutide and weight loss) and at week 44 (assessment of the weight-loss after discontinuation of liraglutide) the patients are assessed by physical examination, carbon monoxide (CO) diffusion test, pulmonary function test, biomarkers of inflammation (CRP, interleucine-6 (IL-6), monocyte chemitactic protein-1 (MCP-1)), Fluorodeoxyglucose (FDG)/PET-CT scan of the lungs, 6-minute walking test, respiratory polygraphy and validated questionnaires including basic dyspnea index, transition dyspnea index, COPD Assessment Test (CAT)-score, short-form-36 (SF-36) and Epworth Sleepiness Score.

DETAILED DESCRIPTION:
COPD is a common disease characterized by pulmonary inflammation, reduced pulmonary capacity, reduced physical activity and quality of life. Obesity is likewise a common disease characterized by inflammation, reduced physical activity and quality of life. Targeting both obesity and inflammation may turn out beneficial for patients with COPD and obesity, and this study explore the possibility to reverse a vicious cycle of COPD, lack of physical activity and obesity. The primary objective of the study is to evaluate the effect of Liraglutide 3mg in patients with COPD on patient reported outcomes as measured by the Transition Dyspnea Index. The hypothesis is that Liraglutide 3mg exerts beneficial effects on measures of pulmonary function and quality of life in overweight patients with COPD by reducing body weight and reducing inflammatory activity.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities
2. COPD as defined by FEV1/FVC<70% after maximal broncho-dilatation and in accordance with the Gold guidelines 2017 (25)
3. Previous smoking of ≥ 20 pack-years
4. Overweight defined as BMI > 27 kg/m2
5. Age 30 - 75 years
6. Women of childbearing potential must use a safe anti-contraceptive method

Exclusion Criteria:

1. Chronic treatment with systemic steroids (inhalation steroids allowed)
2. Current smokers
3. Diabetes mellitus type 1 and type 2 as defined by current or previous treatment with antidiabetic medications of any kind or HbA1c ≥ 48mmol/mol
4. Severe hepatic disease (Alanine transferase > 3 x UNL)
5. Severe impaired renal function (eGFR < 30ml/min)
6. Congestive heart disease New York Heart Association (NYHA) class 3-4
7. History of acute or chronic pancreatitis
8. History of cholecystitis or cholecystolithiasis
9. Pregnant or breastfeeding women
10. Known bronchial asthma or interstitial lung disease
11. Family history of multiple endocrine neoplasia type 2 (MEN2) or medullary thyroid carcinoma
12. Large goiter or plasma-calcitonin > 50ng/ml

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Transition Dyspnea Index (TDI) | 40 weeks
  The primary objective is to evaluate the effect of Liraglutide 3mg on Transition Dyspnea Index (TDI) after 40 weeks of treatment in subjects with COPD and overweight (BMI>27 kg/m2). A positive value indicates less dyspnea during specified activities

SECONDARY OUTCOMES:
6 minutes walking test | 44 weeks
  Walking distance during a 6-minutes walking test
Diffusion capacity of the lung for carbon monoxide (DLCO) | 44 weeks
  Pulmonary Diffusion Capacity measured by Carbon Monoxide (CO) diffusion capacity test
FEV1/FVC | 44 weeks
  Forced expiratory volume in first second (FEV1)/forced vital capacity (FVC)
Total lung capacity (TLC) | 44 weeks
  Total lung capacity
Residual volume (RV) | 44 weeks
  Residual volume
CAT-score | 44 weeks
  Chronic Obstructive Pulmonary Disease assessment test, a measure of COPD impact on every day life, total score ranges 0-25, a higher score indicates more symptoms
SF-36 | 44 weeks
  Short Form (36) Health Survey, which is a Quality of life questionnaire score, subscale scores are calculated according to the SF-36 manual
CRP | 44 weeks
  Inflammation marker, C-reactive protein, higher value indicates more inflammation
IL-6 | 44 weeks
  Inflammation marker, Interleukine 6, higher values indicates more inflammation
MCP-1 | 44 weeks
  Inflammation marker, Monocyte Chemoattractant Protein-1, higher value indicates more inflammation
Maximal standard uptake value (SUV max) | Twice over 44 weeks
  Maximal standard uptake value as measure by FDG-PET/CT scan of the lungs, a higher value indicates more inflammation
Mean standard uptake value (SUV mean) | Twice over 44 weeks
  Mean standard uptake value as measured by FDG-PET/CT scan of the lungs, a higher value indicates more inflammation
Total lesion glycolysis (TLG) | Twice over 44 weeks
  Total lesion glycolysis as measured by FDG-PET/CT, a higher value indicates more inflammation
Body weight | 44 weeks
  Changes in body weight
Number of COPD exacerbations | 44 weeks
  Mild-moderate exacerbations: Treatment with antibiotics or/and oral prednisolone and Moderate-severe exacerbations: Hospitalization due to pulmonary symptoms.
Changes in use of bronchodilator drugs and anti-inflammatory drugs | 44 weeks
  Defined by an increase in beta2agonists of more than 20 % per week and a change of more than 20 % of dose of anti-inflammatory drugs respectively.
Apnea/hypopnea index (AHI) | Twice during 44 weeks
  Apnea/hypopnea index, higher value indicates more apnea/hypopnea episodes
Oxygen desaturation index (ODI) | Twice during 44 weeks
  Oxygen desaturation index, higher values indicate more episodes of desaturation
Epworth score | Twice during 44 weeks
  Epworth sleepiness scale questionnaire, total score is calculated, 0-9: Normal, 10-15: mild to moderate sleep apnea, 16 or more indicate severe sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Claus B Juhl, MD PhD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (2):
- Denmark (2):
  - Hospital of South West Jutland, Esbjerg
  - Lillebaelt Hospital, Vejle

REFERENCES:
- [Derived] Dogan ADA, Christensen TQ, Jensen TT, Juhl CB, Hilberg O, Bladbjerg EM, Hess S. FDG-PET/CT-based respiration-gated lung segmentation and quantification of lung inflammation in COPD patients. BMC Res Notes. 2024 Jun 20;17(1):170. doi: 10.1186/s13104-024-06820-w. PMID 38902794